CLINICAL TRIAL: NCT06145360
Title: Effectivity of Empagliflozin Addition to Insulin and Oral Antidiabetic Medication (OAD) Regimen in Poorly Controlled Type 2 Diabetes
Brief Title: Evaluating the Efficacy and Safety of Empagliflozin Addition to Insulin and Oral Antidiabetic Medication (OAD) Regimen in Poorly Controlled Type 2 Diabetes and Obese Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Collaborators: Horizon Pharmaceutical Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 00003
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-11

CONDITIONS: Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Hypoglycemic Agents; Empagliflozin
Keywords: Insulin Resistance; Type 2 Diabetes; Overweight; Add-on therapy; Glycemic control
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Insulin Resistance; Overweight | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: An adaptive research design was judiciously employed to navigate the complexities of this research. Leveraging a secondary dataset, the study engaged data from registered diabetic patients who had been consistently monitored by SINA over the past six months. These existing datasets formed the foundation for analysis, enabling informed decision-making. Based on rigorous analytical evaluations, a standardized treatment protocol was established, with patients prescribed Empagliflozin 10mg for a duration of three months
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 10mg (Experimental): Group A: Empagliflozin 10 mg once daily with antidiabetic drugs
  Interventions: Drug: Empagliflozin 10 MG
- regimen of Insulin+Metformin+DPP4 inhibitor (DPP4I) (Active Comparator): Group B: usual care group [Insulin+Metformin+DPP4 inhibitor (DPP4I)] but without Empagliflozin with adjustment of therapy as the standard of care.
  Interventions: Drug: Insulin+Metformin+DPP4 inhibitor (DPP4I)

INTERVENTIONS:
Drug: Empagliflozin 10 MG — the impact of incorporating Empagliflozin, an oral sodium-glucose co-transporter 2 (SGLT2) inhibitor, into the existing therapeutic regimen of Insulin+Metformin+DPP4 inhibitor (DPP4I) in poorly controlled type 2 diabetes mellitus (T2DM
  Other Names: EMPAA
  Arms: Empagliflozin 10mg
Drug: Insulin+Metformin+DPP4 inhibitor (DPP4I) — Group B: usual care group but without Empagliflozin with adjustment of therapy as the standard of care
  Arms: regimen of Insulin+Metformin+DPP4 inhibitor (DPP4I)

SUMMARY:
The primary aim of this study is to assess the impact of incorporating Empagliflozin, an oral sodium-glucose co-transporter 2 (SGLT2) inhibitor, into the existing therapeutic regimen of Insulin+Metformin+Dipeptidyl peptidase 4 (DPP-4) inhibitors in poorly controlled type 2 diabetes mellitus (T2DM) patients. The study seeks to evaluate its effect on achieving glycemic goals in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 years or older, diagnosed with Type 2 Diabetes Mellitus,
* Specifically, individuals with a documented HbA1c level equal to or exceeding 8.5% over the course of the last six months or more are considered eligible candidates.
* these patients should currently be undergoing treatment involving a combination of Insulin and either Metformin or Sitagliptin.

Exclusion Criteria:

* Patients with a history of recurrent urinary tract infections
* those who are currently pregnant are excluded from participation in the study.
* patients with an estimated Glomerular Filtration Rate (eGFR) exceeding 40 ml/min/1.73m²,
* Furthermore, individuals with other concurrent medical conditions, and those who are unable to provide informed consent for the study, have also been excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants achieved HbA1c level i.e. <7% | 12 weeks
  The foremost objective is to determine whether the addition of Empagliflozin to the current treatment regimen leads to a significant improvement in glycemic control i.e. glycated haemoglobin less than 7% among poorly controlled T2DM patients in three months of treatment

SECONDARY OUTCOMES:
Weight in Kg | 12 weeks
  Number of participants reduces weight in Kg during the therapy or mean reduction in weight overtime
BMI in kg/m2 | 12 weeks
  Number of participants reduces BMI kg/m2 or mean reduction in BMI overtime
systolic blood pressure and diastolic blood pressure | 12 weeks
  systolic blood pressure and diastolic blood pressure measure in mmHg during the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hina Sharif, Pharm-D,MSPH, Principal Investigator — SINA Health Education & Welfare Trust
Locations (1):
- SINA Shireen Jinnah colony, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No